CLINICAL TRIAL: NCT01930578
Title: Bioimpedance Spectroscopy in Humans During Acute Fluid Volume Expansion With Different Crystalloid Solutions
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The Hospital for Sick Children (Other)
Responsible Party: Principal Investigator, Dr. Paul Pencharz, Emeritus Scientist, The Hospital for Sick Children
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: 1000011897
Record Dates: First submitted 2013-07-26; First posted 2013-08-29 (Estimated); Last update posted 2018-01-09 (Actual); Status verified 2018-01

CONDITIONS: HEALTHY
Keywords: bioimpedance analysis; spectroscopy; electrolyte sodium bromide; extracellular water
MeSH Terms: interventions — Therapeutics; Saline Solution

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Treatment with 0.9% normal saline (Experimental): 1 litre of normal saline infused over minutes and BIS performed at baseline, and 5 minute intervals during infusion, then 5 minute interval readings for 15 minutes after the stop of the infusion.
  Interventions: Other: Treatment with 0.9% normal saline; Other: Treatment with D5+ 0.45 saline; Other: Treatment with D5
- Treatment with D5, 0.45 saline (Experimental): 1 litre of D5, 0.45 saline infused over minutes and BIS performed at baseline, and 5 minute intervals during infusion, then 5 minute interval readings for 15 minutes after the stop of the infusion.
  Interventions: Other: Treatment with 0.9% normal saline; Other: Treatment with D5+ 0.45 saline; Other: Treatment with D5
- Treatment with D5 (Experimental): 1 litre of D5 infused over minutes and BIS performed at baseline, and 5 minute intervals during infusion, then 5 minute interval readings for 15 minutes after the stop of the infusion.
  Interventions: Other: Treatment with 0.9% normal saline; Other: Treatment with D5+ 0.45 saline; Other: Treatment with D5

INTERVENTIONS:
Other: Treatment with 0.9% normal saline — An oral dose of 0.33ml/kg of 10% Sodium Bromide solution at each of 3 study visits. Each dose of Sodium Bromide will be mixed with an equivalent volume; 1:1 of sterile water before oral intake.
  An IV infusion of (1) 0.9% saline, (2) 5% Dextrose or (3) 3.3% Dextrose and 0.3% saline will be given at a rate of 1 liter over an hour in a randomized crossover design.
Other: Treatment with D5+ 0.45 saline — An oral dose of 0.33ml/kg of 10% Sodium Bromide solution at each of 3 study visits. Each dose of Sodium Bromide will be mixed with an equivalent volume; 1:1 of sterile water before oral intake.
  An IV infusion of (1) 0.9% saline, (2) 5% Dextrose or (3) 3.3% Dextrose and 0.3% saline will be given at a rate of 1 liter over an hour in a randomized crossover design.
Other: Treatment with D5 — An oral dose of 0.33ml/kg of 10% Sodium Bromide solution at each of 3 study visits. Each dose of Sodium Bromide will be mixed with an equivalent volume; 1:1 of sterile water before oral intake.
  An IV infusion of (1) 0.9% saline, (2) 5% Dextrose or (3) 3.3% Dextrose and 0.3% saline will be given at a rate of 1 liter over an hour in a randomized crossover design.

SUMMARY:
The objective of the study is to identify a pattern of bioimpedance in humans during acute food changes. As a part of this study the investigators will be administering sodium bromide in oder to measure extracellular water via the bromide dilution technique.

DETAILED DESCRIPTION:
The resistance of the human body to the flow of alternating current is thought to be related to the volume of fluid within the body. The acute change in fluid status of the human body alters the body resistance. This change can be measured accurately with bioelectrical impedance and previous experiments confirmed this observation. However, previous experiments using a piglet model and subsequently humans, suggested that the changes observed is a result of changes in salt instead of body water.

An experiment has shown that bioimpedance analysis (BIA) was able to detect changes in total body resistance when different electrolyte solutions were infused. The changes in resistance were related to changes in osmolarity and electro-ionic state, not to volume of water infused. Therefore, BIA measures principally the electro-ionic state. Thus a measurement of fluid volume can be indirectly obtained from BIA. However, in the non-steady state such as acute fluid volume expansion, the measurement of water volume cannot be performed accurately.

In this study, we will be administering sodium bromide in oder to measure extracellular water via the bromide solution technique. Despite the interesting observations, the human study described above was underpowered. Therefore, we aim to validate the observations that have been previously made through carrying out an appropriately powered study with an adequate sample size to validate the observations noted.

ELIGIBILITY:
Inclusion Criteria:

* Age > 18 years
* Otherwise healthy with no medical history of: cardiac disease, renal disease, chronic liver disease, diabetes, or lymphedema

Exclusion Criteria:

* Allergy to bromide
* Breast feeding mothers
* Pregnancy
* Heart failure
* Presence of a pace maker
* Renal failure
* Any contraindication to fluid bolus
* Recent or continued exposure to bromide containing drugs

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2008-05; Primary Completion 2008-06 (Actual); Study Completion 2008-06 (Actual)

PRIMARY OUTCOMES:
Pattern of bioimpedance in humans during acute food changes. | 3 hours
Bioimpedance spectroscopy in humans | 3 hours
  change in bioimpedance spectroscopy (MHz)in humans during acute fluid expansion as a result of administration of different intravenous crystalloid solutions

CONTACTS AND LOCATIONS:
Overall Officials: Paul Pencharz, MD, Principal Investigator — The Hospital for Sick Children
Locations (1):
- The Hospital for Sick Children, Toronto, Ontario, Canada

REFERENCES:
- [Background] Yap J, Rafii M, Azcue M, Pencharz P. Effect of Intravenous Infusion Solutions on Bioelectrical Impedance Spectroscopy. JPEN J Parenter Enteral Nutr. 2017 May;41(4):641-646. doi: 10.1177/0148607115619598. Epub 2015 Dec 4. PMID 26637229